CLINICAL TRIAL: NCT04683705
Title: Ultrasound Measurement of the Suprascapular Nerve in Asymptomatic and Painful Shoulders
Brief Title: Ultrasound Measurement of the Suprascapular Nerve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20180405RIND
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Shoulder Pain
Keywords: Ultrasonography; Rotator cuff; Suprascapular Nerve; Pain
MeSH Terms: conditions — Shoulder Pain; Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients without shoulder pain: This was a cross-sectional study investigating suprascapular nerves in the asymptomatic shoulders of participants. All the participants were required to ambulate independently, have normal cognitive function and complete the given questionnaires. The group included at least 60 participants.
  Interventions: Diagnostic Test: Ultrasound
- patients with shoulder pain: This was a cross-sectional study investigating suprascapular nerves in the painful shoulders of participants. All the participants were required to ambulate independently, have normal cognitive function and complete the given questionnaires. The group included at least 60 participants.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — 1. High-resolution ultrasound evaluation of the shoulder region to recognize the biceps tendon, subscapularis tendon, supraspinatus tendon, and infraspinatus tendon.
  2. High-resolution ultrasound evaluation for the C5, C6 and C7 nerve roots and the suprascapular nerve over the supraclavicular fossa , in the supraspinatus fossa and in the infraspinatus fossa to obtain the nerve cross-sectional image.
  3. Collecting the shoulder pain-related information, including physical examination results (bicipital groove tenderness, Speed test, Yergason's test, Empty can test, Neer test, Hawkins-Kennedy test and painful arc test) and status of disability using Shoulder Pain and Disability Index (SPADI).

SUMMARY:
Suprascapular nerve is the first nerve that branches from the upper trunk of brachial plexus. It receives signals transmitted from the fifth and sixth cervical root. The clinical importance of suprascapular nerve is mainly based on its distribution of 70% sensory innervation to the glenohumeral joint. After divided from the upper trunk, the suprascapular nerve goes laterally and posteriorly. First, it passes underneath omohyoid muscle, and then goes through the suprascapular notch and into the suprascapular fossa. At suprascapular fossa, the suprascapular nerve is just below supraspinatus muscle. If there are some problems inside the supraspinatus muscle, the suprascapular nerve below it could be compromised. After suprascapular nerve passes suprascapular fossa, it will cross spinoglenoid notch, then go into infraspinatus fossa and innervates infraspinatus muscle. Based on the important distribution of suprascapular nerve to the sensory and motor function of shoulder joint, it has great benefits to understand its normal and abnormal sonographic images in order to diagnose refractory shoulder pain cases. Although there are some studies trying to measure the size of suprascapular nerve, most of them are limited in its location at the supraspinatus fossa. Also, they do not take factors into consideration, such as the subject's sex, body index, orientation and if shoulder pain or not at that point. In conclusion, our study is aimed to explore the difference of the suprascapular nerves between the participants with and without shoulder pain and to investigate potential factors that may influence the nerve's size using high-resolution ultrasound.

DETAILED DESCRIPTION:
Introduction:

Shoulder pain arises to be one of the most common musculoskeletal complaints. The mechanism of an increased risk of painful shoulders is multifactorial and the role of the suprascapular nerve in development and management of shoulder pain has been highlighted recently. In recent years, high resolution ultrasound has been widely applied on evaluation of entrapment neuropathy, and its reliability on assessing the cross-sectional area of suprascapular nerves has been validated. As the suprascapular nerve is crucial for conducting shoulder motion and sensation, it is of clinical importance to measure the size of suprascapular nerve. Our study is aimed to explore the difference of the suprascapular nerves between the participants with and without shoulder pain and to investigate potential factors that may influence the nerve's size using high-resolution ultrasound.

Material and methods:

Study design:

This was a cross-sectional study investigating suprascapular nerves in the asymptomatic and painful shoulders of participants. All the participants were required to ambulate independently, have normal cognitive function and complete the given questionnaires. Both groups included at least 60 participants.

Detail of the investigation

1. High-resolution ultrasound evaluation of the shoulder region to recognize the biceps tendon, subscapularis tendon, supraspinatus tendon, and infraspinatus tendon.
2. High-resolution ultrasound evaluation for the C5, C6 and C7 nerve roots and the suprascapular nerve over the supraclavicular fossa, in the supraspinatus fossa and in the infraspinatus fossa to obtain the nerve cross-sectional image.
3. Collecting the shoulder pain-related information, including physical examination results (bicipital groove tenderness, Speed test, Yergason's test, Empty can test, Neer test, Hawkins-Kennedy test and painful arc test) and status of disability using Shoulder Pain and Disability Index (SPADI).
4. The measurements of the nerve cross-sectional area were conducted by another specialist with the image processing software (Image J). For the most proximal section of the suprascapular nerve, the cross-section of the nerve fascicles inside the hyperechoic epineurium were measured. In the segment over the supraspinatus and infraspinatus fossae, the whole nerve's cross-section including its epineurium were measured.
5. The identification for the images of the rotator cuff lesions or biceps tendon lesions were conducted by another specialist.
6. Comparison of age, body height, body weight, and CSA across various age and sex groups were conducted.

Statistical analysis:

1. Continuous variables: Mann Whitney u test
2. Categorical variables: Chi-square test

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 20 year old). All the participants were those visiting the department of physical medicine and rehabilitation for musculoskeletal complaints.

Exclusion Criteria:

* History of malignancy
* Uncontrolled medical conditions (like systemic rheumatic disease, including rheumatic arthritis and ankylosing spondylitis).
* Previous major trauma or surgeries, and suprascapular nerve block on either side of the shoulders within the three months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants: Adult patients (≥ 20 year old). All the participants were those visiting the department of physical medicine and rehabilitation for musculoskeletal complaints.
  Control : Healthy asymptomatic volunteers, adult subjects (≥20 year old)
  Exclusion criteria:
  The exclusion criteria included history of malignancy, uncontrolled medical conditions (like systemic rheumatic disease, including rheumatic arthritis and ankylosing spondylitis), previous major trauma or surgeries, and suprascapular nerve block on either side of the shoulders within the three months.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Nerve cross-sectional area | During/at recruitment.
  The measurements of the nerve cross-sectional area were conducted by another specialist with the image processing software (Image J). For the most proximal section of the suprascapular nerve, the cross-section of the nerve fascicles inside the hyperechoic epineurium were measured. In the segment over the supraspinatus and infraspinatus fossae, the whole nerve's cross-section including its epineurium were measured.
The Chinese version of the Shoulder Pain and Disability Index (SPADI) tool | During/at recruitment.
  The Chinese version of the Shoulder Pain and Disability Index (SPADI) tool. The SPADI tool consisted of 13 questions categorized in two domains: pain and disability. They were instructed to indicate the level of influence on a 10 cm visual analogue scale for each question with a rating from 0 (no pain or no difficulty) to 10 (worst pain or extreme difficulty). The scores from the pain and functional domains were averaged to generate the total score of SPADI, with a highest value of 100 points.
Visual analogue scale | During/at recruitment.
  The pain scale to evaluate pain, from 0 to 10. The lower means less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Vin Chang, MD,PhD, Study Chair — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital, Bei-Hu Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No